CLINICAL TRIAL: NCT04435405
Title: Micro-Analysis of Processes in a Group Music Therapy for People Living With Mental Health Conditions in the Community: a Quantitative Single-Cases Study
Brief Title: Micro-Analysis of Processes in a Group Music Therapy for People Living With MHC in the Community
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: 149/20
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Mental Health Disorders
Keywords: Community music therapy; Video micro-analysis
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Video microanalisys: Video footage analysis of group and individual behavioral processes.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — video footage analysis of group and individual behavioral processes.

SUMMARY:
People with mental health conditions (MHC) often face significant barriers in obtaining personal valued social roles and feeling a sense of belonging to their community. With the growing emphasis on community integration, and the fact that the vast majority of people with MHC live in the community, there is an effort to develop interventions and services which focus on recovery, wellbeing, and community integration, to reclaim "right to a safe, dignified, and personal and gratifying life in the community despite his or her psychiatric condition" (Davidson, Tondora, Lawless, O'Connell, & Rowe, 2009, p.11).Music therapy (MT) has been practiced for many decades with growing evidence for its effectiveness in different populations, including people with MHC. Music has pivotal influences on socialization and in building inter-personal skills and has the potential to be effective as a community-based therapeutic approach in bringing people together in a shared experience, an important step towards integration back to the community. MT encourages verbal and non-verbal interactions and offers opportunity to practice interpersonal skills, build relationships and peruse common goals.

The proposed study has a potential to shed additional light on the processes of recovery in people living in the community with MHC who are participating in group CoMT. Although the study will pinpoint to the domains where MT was mostly studied before (social skills, group cohesion and emotional expression), it is unique in two main aspects:

1. Majority of previous MT studies on people with MHC were testing short-term MT interventions in in-patient brief settings. This has limited significance in understanding the generalization of MT into everyday life and promoting wellbeing. In the proposed study, on the other hand, I will try to evaluate the significance of recovery-oriented long-term group CoMT in the community, where most people live, focusing on behavioral domains where MT is expected to benefit most: The client's social skills development, group cohesion and emotional expression (affect improvement).
2. This study, to my knowledge, is the first that is based on longitudinal quantitative micro-analysis of filmed video sessions. This approach bypasses the participants subjective reaction to a qualitative interview (which by itself is important) allowing an additional un-biased angle of observation on the interaction process (assuming that the participants may ignore the presence of the video camera over time).

DETAILED DESCRIPTION:
This was an exploratory, retrospective, quantitative, longitudinal single-cases study.

The study was designed to observe the development of different behavioral, emotional, social and musical domains as well as the development of group cohesion during 9 months of weekly group CoMT. These behaviors were chosen since they can serve as indicators for satisfying social recovery and wellbeing (Wilson et al., 2008; Tew et al., 2012; Solli et al.,2013;Jetten et al., 2014 ; Solli, 2015), can build up gradually through group meetings, and can simply be observed and quantified.

For this, video recorded sessions were quantitively micro-analyzed by 2 scales: one that tests individual participants performance, the second tests the group performance as a whole. The scales score several behavioral domains, focusing on social skills, affect and group cohesion.

Ethical considerations: The study protocol and informed consent form (ICF) were approved, prior to data collection, by the ethics committee for the evaluation of research with human subjects of the faculty of social welfare & health sciences, Haifa University, Israel. Participants were informed on the study, its purposes, design, and conduct both orally and by explanation leaflet. Following this, all participants signed an ICF. Participant confidentiality was maintained at all times. Confidential private data was not exposed in the video recordings.

Data, including the video films, were stored and handled securely, and were destroyed upon study completion.

The study was registered in ClinicalTrials.gov (XXX). The data collected in this study in available as a supplementary document to this manuscript.

Participants and setting The study involved eight adult individuals (20-65 years old) of both genders, who are long term service-users with MHC (schizophrenia and schizoaffective disorders). The participants took part in a weekly community music therapy group in "Enosh" community center. The declared goal of this CoMT group was defined as a music therapy project based on individual and group work, that invites the participants to share and express emotional and daily life experiences through singing, improvising, playing instruments and creating original songs.

All group participants were eligible to be included to the study. The participants had a strong interest in music, although it was not an inclusion criterion. The participants had no previous music experience. Only participants whose behavior was fully captured in all video-recordings were included in the individual behavior analysis, thus four out of the eight individuals fulfilled this criterion and their behaviors were analyzed.

The CoMT sessions were co-facilitated by a certified music therapist, trained for community music therapy practice, and a psychiatrist. Both the music therapist and the psychiatrist received ongoing advanced training from a senior music therapist experienced in the field of CoMT.

The CoMT group followed a pre-defined protocol and the extent to which the delivery of the intervention adheres to the protocol was monitored. This was done on two levels: individual and group. The music therapist performed weekly individual sessions, which included original song-writing based on the preferences of the participant, to explore if the CoMT meets the participant's goals, needs and expectations. On the group level, a wide variety of musical engagement were involved, including free improvisations, singing from song-books and the participant's original songs, and playing instruments. In addition, periodic discussions were held after the sessions to explore if the group goals were met and changes were applied accordingly.

Data analysis method Longitudinal video micro-analysis was performed on the video films to answer the main research question: whether recovery-oriented long-term group CoMT be beneficial in social skills development, group cohesion and affect improvement. According to Wigram, and Wosch (2007), video microanalysis is a comprehensive and a powerful tool when investigating aspects related to interaction and communication. Assessment of video films have successfully been used before to explore the long-term effects of psychotherapeutic interventions in people with MHC (Isbell, Thorne and Lawler 1992; Lee and McFerren 2015; Wang, Yang and Yu 2018).

Five MT sessions, out of 30 filmed during the course of group music therapy were selected for the study: baseline (at the beginning of the course), after two, four and five months and at the end of the course (9 months).

Video recording micro-analysis was based on two scales: the first for individual participant assessment - Individual Behavior Observation Categorization Scale, (Mercadal-Brotons,2014) the second for group assessment - Group Environmental Scale (Isbell, Thorne and Lawler 1992; Lee and McFerren 2015; Wang, Yang and Yu 2018).

Assessment was carried out by three blinded raters (blinded to the timepoint of the filmed session) for the group analysis and by one blinded rater for the individual analysis. In order to reduce inter-rater variability, the raters were trained on the use of the group analysis scale in analyzing videos (which were not from those intended for the study evaluation). The training continued until raters consent was achieved.

The study was planned with a small sample size, underpowered to conclusively confirm or disconfirm beneficial effects of CoMT in this group of people, but adequate to probe for signal of potential benefit for future large-scale confirmatory study design.

Statistical analysis was carried out by the F test with N=4 (# of time points), force zero intercept, 3 degrees of freedom to identify if there was statistically significant difference over time. This statistical test evaluates the change between each time point to the baseline.

The Scales

Scale to assess individual performance

The Individual Behavior Observation Categorization Scale (IBOC scale):

The IBOC scale is an appraisal method that measures behavior against levels of performance and also measures the frequency with which the behaviors occur. It is commonly used in the medical arena, as well as job performance in school and work environments, and other uses. In brief, the instruments of IBOC is either ordinal scale questionnaire and/or counting the frequency of the tested behavior. The scale was successfully used before to analyze videos of MT sessions in dementia patients, and music participation behaviors were adopted into the scale (Sole et al., 2014).

The scale tests 5 behavioral categories which are simple to quantify in a video film (Mercadal-brotons,2014). Each of these categories is further divided into sub-categories: Verbalization, Physical contact, Visual contact (gaze), Active participation in music activities, and Emotions/facial affect and body expressions.

The rater quantified the number of specific events that the tested individuals exhibited, for example, how many times in the session the individual had visual contacts with other participants. A behavior category score is the sum of all the sub-categories of the score. The whole session lasts 1 hours and the assessment was carried out between minute 23-46 (overall 23 minutes of each session). This time frame was suggested by the music therapist as it represents the time frame were the musical activity is the most pronounced during the meeting.

The IBOC scale is highly relevant to the study as it focuses on the domains of social skills and group cohesion, participation in music activity, and affect (emotional expression):

* Social skills and group cohesion = Verbalization, Physical contact, Visual contact (gaze) and Active participation in music activities.
* Participation in music activity = to assess the degree of engagement in singing, playing instruments, music listening & improvisation.
* Affect = Emotional expression.

Repeating the micro-analysis in 5 time points enabled a longitudinal analysis of the CoMT process on the chosen participants.. A test for regression slope (the F test) was used to assess whether a trend of improvement is demonstrated per category per participant over time. The H0 assumed no change in score.

Scale to assess group performance Group Environmental Scale (GES) In brief, the GES offers a quantitative method for assessing intervention support groups (Moos RH 1994). The GES has (1) psychometrically established reliability, factor structure, content, and construct validity (2) has generic applicability to different types of groups from different settings, (3) has subscales theoretically matching most support group objectives and expands into "leader" and "systems maintenance" dimensions, and (4) is brief, taking short time to complete 90 true/false items on an answer form, with additive responses easily converted into a 9-point interval scale for standardized scoring. GES was originally designed to be rated by group members. To make it suitable for external rating, we slightly altered the wording of the questions without changing their meanings.

GES was used before to analyze different group interventions and group environments including in mental health patients (Lavoie 1981; Isbell, Thorne, Ph, Lawler, & Ed, 1992).

GES evaluates 10 "group environment" subscales: Cohesion, Leader (therapist) support, Expressiveness, Independence, Task orientation, Self-discover, Anger and aggression, Order and organization, Leader control, and Innovation.

Each subclass has 9 Yes/No questions (total of 90 questions). The rater watches the video and at the end answers the 90 questions. "Yes"- scores 1, "No" - score 0, and each subclass score is the total score of its 9 questions.

The GES is highly relevant to the study as it focuses on group cohesion domains as follows:

* Relationship = Cohesion, leader support, Expressiveness.
* Personal Growth = Independence, Task orientation, Self-discovery, ( - ) Aggression.
* System maintenance and change = Order and organization, Leader control, Innovation.

Repeating the micro-analysis in the different time points enabled a longitudinal analysis of the CoMT process on the group.

The F test for regression slope was used to assess whether a trend of improvement is demonstrated per domain over time. The H0 assumes no change in score.

ELIGIBILITY:
Inclusion Criteria:

* All group participants are eligible to be included to the study

Exclusion Criteria:

* Only participants whose behavior is fully captured in all video-recordings are to be included in the individual behavior analysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves adult individuals , who are long term service-users with Mental Health Conditions . The participants take part in a weekly community music therapy group in community center.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Change in the score of the Group Environmental Scale within 9 months | 9 months
  Social skills, group cohesion and affect improvement change from baseline to nine months is evaluated by the Group Environmental Scale. The minimal score is "0" and the maximal score is "90" while the higher score indicates a better outcome.

SECONDARY OUTCOMES:
Change in the score of the active participation in musical activities section of the Individual Behavior Observation Categorization Scale within 9 months. | 9 months
  Musical activities improvement change from baseline to nine months is evaluated by the musical activities section of the Individual Behavior Observation Categorization Scale. The score is based on counting the frequency of the activities with a minimal frequency of "0". The higher the score, the better outcome.
Change in the score of the Individual Behavior Observation Categorization Scale within 9 months. | 9 months
  The improvement change of social skills and affect from baseline to nine months is evaluated by the total score of the Individual Behavior Observation Categorization Scale. The score is based on counting the frequency of the activities with a minimal frequency of "0". The higher the score, the better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: starting 6 months after publication